CLINICAL TRIAL: NCT07055997
Title: The Effectiveness of Robotic-assisted Navigation System for Preoperative Lung Nodule Localization: a Prospective, Single-center, Non-inferiority Clinical Study
Brief Title: Robotic-Assisted Navigation for Lung Nodule Localization: A Non-Inferiority Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ES-2024-129-02
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Lung Nodules; Lung Cancer (Diagnosis); Robotic-Assisted Navigation System
Keywords: Robotic-assisted; lung nodule; preoperative localization; video-assisted thoracoscopic surgery (VATS); non-inferiority study
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freehand group (Active Comparator): Manual CT-guided percutaneous needle localization of pulmonary nodules
  Interventions: Procedure: Manual needle localization
- Robotic group (Experimental): Robotic-assisted CT-guided percutaneous needle localization of pulmonary nodules
  Interventions: Device: Robotic-assisted needle localization

INTERVENTIONS:
Device: Robotic-assisted needle localization — Robot-assisted needle localization involves the use of a robotic system to assist with the percutaneous localization of pulmonary nodules under CT guidance. The robotic system provides real-time navigation and increased precision during needle placement, reducing the variability in positioning and improving the accuracy of localization. The system offers automatic adjustments to the needle's trajectory, minimizing the need for manual corrections, and potentially reducing the number of CT scans required. This method is designed to enhance the overall localization success rate and reduce complications associated with traditional manual techniques.
  Arms: Robotic group
Procedure: Manual needle localization — Manual needle localization involves the traditional technique of percutaneous localization of pulmonary nodules under CT guidance without the assistance of robotic systems. The procedure is performed by the physician manually guiding the needle based on real-time CT imaging. The physician adjusts the needle position based on visual cues from the CT scan, which may require multiple attempts for accurate localization.
  Arms: Freehand group

SUMMARY:
This study compares robotic-assisted navigation and manual CT-guided needle localization for lung nodules under 20 mm. It aims to evaluate localization success, procedure duration, CT scans, and complication rates.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-inferiority clinical study designed to evaluate the effectiveness of a robotic-assisted navigation system for lung nodule localization compared to traditional manual CT-guided needle localization. The study will be conducted between June 2024 and December 2024, involving 100 patients with lung nodules smaller than 20 mm in diameter. Participants will be randomly assigned to receive either CT-guided manual needle localization or robotic-assisted needle localization. The primary outcome measure will be the localization success rate, defined as the ability to accurately locate the nodule and guide the needle to the target site for biopsy or surgery. Secondary outcome measures will include procedural duration, the number of CT scans required, total dose-length product (DLP), first-pass success rate, localization success within a single needle adjustment, and complication rate.

ELIGIBILITY:
Inclusion Criteria:

(Ⅰ) isolated pulmonary nodules with a maximum diameter of less than 20 mm; (Ⅱ) the presence of pure ground-glass opacity (GGO) or mixed GGO (solid to tumor ratio < 0.5) on CT with clinical or radiological suspicion of malignancy; (Ⅲ) patient with a peripheral nodule, located in the outer third of the lung parenchyma, with its edge situated at least 5 mm away from the pleural surface; (Ⅳ) Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-1, indicating suitability for surgical intervention.

Exclusion Criteria:

(Ⅰ) nodule location obstructed by the scapula, precluding needle access; (Ⅱ) proximity of the nodule to major blood vessels, defined as within 2 cm; (Ⅲ) requirement for localization of multiple pulmonary nodules.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Localization Success Rate | Immediately after needle localization and before surgery
  The accuracy of nodule localization was designated as the primary outcome of the study. Successful localization was defined as a distance of less than 10 mm between the needle tip and the center of the nodule, with no displacement of the localization device between localization and surgery.

SECONDARY OUTCOMES:
Procedure Duration | From patient positioning on the CT scanner to confirmation of successful needle insertion via final CT scan
  Procedure duration was calculated from the time the patient was positioned on the CT scanner to the confirmation of successful needle insertion via the final CT scan.
Number of CT Scans Required for Localization | During the localization procedure
  The number of CT scans needed to successfully localize the nodule.
Total Dose-Length Product (DLP) | During the localization procedure
  The total dose-length product (DLP) accumulated during the localization process.
First-pass Success Rate | Immediately after the first needle insertion
  First-pass success was defined as the successful localization of the nodule with the first needle insertion, without requiring any needle adjustment.
Localization Success Rate within One Needle Adjustment | Immediately after one needle adjustment
  The localization success rate within one needle adjustment was defined as successful localization achieved after a single adjustment to the needle's depth or angle following initial misplacement.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated of Guangzhou Medical University, Guangzhou, Guangdong, China